CLINICAL TRIAL: NCT02113020
Title: A Randomized, Double-blind, Single-dose, 4 × 4 Crossover Phase I Study to Examine the Effects of TAK-233 on the Urethral Function in Healthy Female Subjects
Brief Title: A Phase I Clinical Pharmacology Study of TAK-233 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: TAK-233/CPH-003; U1111-1152-9381 (Registry Identifier: WHO)
Record Dates: First submitted 2014-02-21; First posted 2014-04-14 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Clinical Pharmacology

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAK-233 (Experimental): Oral administration
  Interventions: Drug: TAK-233
- Placebo (Placebo Comparator): Oral administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAK-233 — Oral administration of TAK-233
  Arms: TAK-233
Drug: Placebo — Oral admininstration of Placebo
  Arms: Placebo

SUMMARY:
The objective of this clinical trial is to examine the clinical pharmacology properties of TAK-233 in healthy female subjects

DETAILED DESCRIPTION:
The primary objective of this study is to examine the pharmacodynamics and the safety of TAK-233 administered as a single dose in healthy women.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who understand the contents of this clinical trial and who the investigator or sub-investigator consider able to comply with the procedures of the clinical trial
2. Subjects who can sign the informed consent form and can date the form without assistance before starting the procedures of the clinical trial
3. Healthy Japanese women
4. Subjects aged ≥ 20 and ≤ 40 years at the time of consent
5. Subjects with body weight ≥ 45 kg and BMI ≥18.5 and ≤ 25.0 kg/m2 at the time of screening
6. Women of child bearing potential who agree to take specified contraceptive measures regularly from the time of consent until 4 weeks after the end of the last assessment in the fourth treatment period

Exclusion Criteria:

1. Subjects who received TAK-233 within 16 weeks before the start of initial administration
2. Subjects who have previously received TAK-233 during treatment or during participation in another clinical trial
3. Employees of the medical institution conducting this clinical trial and their family/dependents (e.g., husband or wife, parents, children, and siblings), or subjects who may be coerced to agree to participate in the clinical trial
4. Subjects with poorly controlled and clinically significant neurological, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal (including chronic costiveness), urological (including dysuria), autoimmune, endocrine, or psychiatric diseases or other abnormalities which may affect the subject's participation in the clinical trial or results of the clinical trial
5. Subjects with hypersensitivity to TAK-233 related substances, or excipients of these products
6. Subjects whose urine tested positive for drug abuse at screening
7. Subjects with a history of drug abuse (defined as the use of illegal drugs) or alcohol dependence within 52 weeks before the screening assessments, or subjects who are not willing to stop alcohol intake or drug use during their participation in the clinical trial
8. Subjects who need to take prohibited concomitant medications, vitamins, or foods listed in listed in what?
9. Pregnant or lactating women, women expecting to be pregnant before giving consent, during this clinical trial, or within 4 weeks after the completion of this clinical trial, or women who are planning to donate their ova during this period
10. Subjects with currently active cardiovascular diseases, central nervous system diseases, hepatic diseases, hematopoietic diseases, renal failure, metabolic disorders, endocrine disorders, serious allergies, asthma, hypoxemia, hypertension, convulsion, allergic exanthema, or urological disorders (subjects with peptic ulcer, convulsive disorders, or arrhythmia also fall this category)
11. Subjects that have any of the following diseases/surgical interventions that may affect drug absorption: digestive system disorders (malabsorption, esophageal reflux, peptic ulcer, erosive oesophagitis, frequent heartburn (at least once a week), or surgical interventions (e.g., cholecystectomy), or subjects who have had prior history of any of these diseases/surgical interventions within the last 24 weeks
12. Subjects with a history of cancer (excluding subjects whose basal cell carcinoma has been in remission for at least 5 years
13. Subjects that have tested positive for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antigen/antibody, or syphilis serological reaction at screening
14. Subjects who took nicotine-containing products (e.g., cigarette, pipe tobacco, cigar, chewing tobacco, nicotine patch, and nicotine gum) within 28 days before hospitalization
15. Subjects for whom blood collection from peripheral veins is difficult
16. Subjects who donated at least 200 mL of whole blood within 4 weeks before the start of the initial administration, or subjects who donated at least 400 mL of whole blood within 16 weeks before the start of the initial administration
17. Subjects who donated at least 400 mL (in total) of whole blood within 52 weeks before the start of the initial administration
18. Subjects who donated blood components within 2 weeks before the start of the initial administration
19. Subjects with clinically significant abnormalities on the electrocardiogram recorded at screening or hospitalization (Day -1 of the first treatment period)
20. Subjects who had a QTcF interval of > 470 msec or a PR interval of < 120 msec or > 220 msec on the electrocardiogram recorded at screening or hospitalization
21. Subjects with a systolic blood pressure of < 100 mmHg or > 140 mmHg and a diastolic blood pressure of < 60 mmHg or > 90 mmHg at screening or hospitalization
22. Subjects with a heart rate of < 50 bpm or > 90 bpm at screening or hospitalization

22. Subjects unlikely to comply with the protocol, or subjects the investigator or sub-investigator considers ineligible for participation in the clinical trial due to other reasons

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in motor threshold for urethral sphincter contraction. | 0.5 hours post-dose
Change from baseline in motor threshold for urethral sphincter contraction. | 3 hours post-dose
Change from baseline in motor threshold for urethral sphincter contraction. | 6 hours post-dose

SECONDARY OUTCOMES:
Number of participants with adverse events | Up to 28 days
  Treatment emergent adverse events, vital signs, weight, safety ECG, and clinical laboratory tests (hematology, serum chemistry, and urinalysis).

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Takeda
Locations (1):
- Kumamoto, Kumamoto, Japan